CLINICAL TRIAL: NCT07189403
Title: A Phase 1, First-in-human (FIH), Multicenter, Open-label Trial of DS9051b in Participants With Advanced or Metastatic Adrenocortical Carcinoma (ACC) and Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: A Study of DS9051b in Participants With Advanced or Metastatic Adrenocortical Carcinoma and Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS9051-079; 2025-521886-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced or Metastatic Adrenocortical Carcinoma; Metastatic Castration-resistant Prostate Cancer
Keywords: Advanced or metastatic adrenocortical carcinoma; Metastatic castration-resistant prostate cancer
MeSH Terms: conditions — Adrenocortical Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DS9051b (Experimental): Participants with advanced or metastatic adrenocortical carcinoma and metastatic castration-resistant prostate cancer who will receive DS9051b.
  Interventions: Drug: DS9051b

INTERVENTIONS:
Drug: DS9051b — Administered orally

SUMMARY:
This FIH study is designed to assess the safety, tolerability, and preliminary efficacy signals of DS9051b in participants with ACC and mCRPC.

DETAILED DESCRIPTION:
The purpose of the dose escalation part is to determine the maximum tolerated dose (MTD) and recommended dose for expansion (RDE), as well as to establish the safety profile of DS9051b in participants with advanced or metastatic ACC and mCRPC.

ELIGIBILITY:
General Inclusion Criteria for All Participants

1. Sign and date the main ICF, prior to the start of any trial-specific procedures.
2. Adults ≥18 years of age at the time the ICF is signed (Follow local regulatory requirements if the legal age of consent for trial participation is >18 years old)
3. Histologically confirmed diagnosis of ACC or adenocarcinoma of the prostate
4. ECOG PS of 0 or 1 assessed no more than 14 days prior to C1D1. (ECOG PS of 2 due to cancer pain is acceptable)
5. Has adequate organ and bone marrow function as assessed by local laboratory within 14 days prior to C1D1 as defined below. Organ and bone marrow function criteria must also be met when laboratory tests are repeated within 3 days of initiation of trial intervention as appropriate.

   Additional Inclusion Criteria for Participants with mCRPC
6. Treatment with at least 1 line (or more) of ARPI therapy for CSPC or in CRPC for a minimum of 12 weeks (eg, abiraterone, enzalutamide, darolutamide, apalutamide).
7. Treatment with at least 1 line (or more) of chemotherapy, having ineligibility for chemotherapy or refusal of chemotherapy.
8. Documented disease progression by one or more of the following criteria:

   * PSA progression as defined by PCWG3 criteria.
   * Soft tissue disease progression as defined by RECIST 1.1 criteria.
   * Bone disease progression as defined by Prostate Cancer Working Group 3 criteria.

An individual who meets any of the following criteria will be excluded from participation in this trial:

1. History of pituitary gland dysfunction.
2. Active or uncontrolled autoimmune disease requiring systemic treatment.
3. Any medical condition (other than the cancer disease) requiring a dose of concurrent systemic corticosteroid treatment greater than 5 mg of prednisone and/or 100 μg of fludrocortisone per day (or equivalent).
4. Active infection or other medical conditions that would make corticosteroids contraindicated.
5. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated, clinically progressive, symptomatic, or requiring systemic therapy with corticosteroids or anticonvulsants or local therapy (ie, radiotherapy) to control associated symptoms.
6. Uncontrolled or significant cardiovascular disease.
7. History of another primary malignancy (beyond the indication[s] under study) except for:

   * Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of trial intervention and of low potential risk for recurrence.
   * Non-melanoma skin cancer, lentigo maligna, or lentigo maligna melanoma treated with curative intent and without evidence of disease.
   * Carcinoma in situ treated with curative intent and without evidence of disease.
   * Participants with a history of prostate cancer (tumor/node/metastasis stage) of Stage ≤T2cN0M0 without biochemical recurrence or progression and who, in the opinion of the investigator, are not deemed to require active intervention.
8. Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE version 5.0, Grade ≤1 or baseline.
9. Participants who cannot swallow whole DS9051b tablets and/or follow DS9051b administration schedule at protocol-defined frequency due to some reasons (eg, dysphagia etc).
10. Known gastrointestinal disease or gastrointestinal procedure that may interfere with absorption of trial intervention including proton pump inhibitors and antacids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting Dose-limiting Toxicities (DLTs), Treatment-emergent Adverse Events (TEAEs), TEAEs Associated With Treatment Discontinuation, Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESI) - All Patients | Baseline up to 50 months
  AEs will be graded using NCI-CTCAE v5.0. A DLT is defined as any TEAE not attributable to disease or disease-related processes, environmental factors, unrelated trauma, etc. that occurs during the DLT evaluation period (Day 1 to the end of Cycle 1) and is Grade ≥3 with exceptions as further defined. TEAEs are defined as those AEs with start or worsening date during the on-treatment period (from the first dose date of trial intervention to 30 days after the last dose date of trial intervention).

SECONDARY OUTCOMES:
Objective Response by Investigator Assessment in Participants With Advanced or Metastatic Adrenocortical Carcinoma and Metastatic Castration-resistant Prostate Cancer | Baseline up to 50 months
  Objective response is defined as participants with a best overall response of confirmed complete response (CR) or confirmed partial response (PR) as assessed by the investigator per RECIST v1.1 (ACC) or PCWG3 (CRPC). CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Disease Control by Investigator Assessment in Participants With Advanced or Metastatic Adrenocortical Carcinoma and Metastatic Castration-resistant Prostate Cancer | Baseline up to 50 months
  Disease control (DC) is defined as participants with a best overall response of confirmed CR or confirmed PR or SD as assessed by the investigator per RECIST v1.1 (ACC) or PCWG3 (CRPC). CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Clinical Benefit by Investigator Assessment in Participants With Advanced or Metastatic Adrenocortical Carcinoma and Metastatic Castration-resistant Prostate Cancer | Baseline up to 50 months
  Clinical benefit is defined as participants with a best overall response of confirmed CR, confirmed PR, or SD lasting ≥183 days as assessed by the investigator per RECIST v1.1 (ACC) or PCWG3 (CRPC). CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Duration of Response by Investigator Assessment in Participants With Advanced or Metastatic Adrenocortical Carcinoma and Metastatic Castration-resistant Prostate Cancer | From date of initial response (CR or PR) to the earlier date of the first objective documentation of radiographic disease progression (based on investigator assessment per RECIST v1.1) or death due to any cause, up to 50 months
  Duration of response (DoR) in a responding participant is defined as the time (in months) from date of initial response (CR or PR) to the earlier date of the first objective documentation of radiographic disease progression (based on investigator assessment per RECIST v1.1 for ACC patients or PCWG3 for CRPC patients) or death due to any cause. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Progression-free Survival by Investigator Assessment in Participants With Advanced or Metastatic Adrenocortical Carcinoma | From the date of the first administration of trial intervention to the earliest date of the first objective documentation of radiographic disease progression or death due to any cause, up to 50 months
  Progression-free survival is defined as the time from the date of the first administration of trial intervention to the earliest date of the first objective documentation of radiographic disease progression as assessed by the investigator per RECIST v1.1 or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Florida Cancer Specialists, Sarasota, Florida
  - Columbia University, New York, New York
  - Brown University, Providence, Rhode Island
- France (2):
  - IUCT Oncopole, Toulouse
  - Centre Oscar Lambret, Villejuif
- Royal Marsden, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/